CLINICAL TRIAL: NCT06985810
Title: Effects of Accentuated Eccentric Loading Versus Flywheel Exercises on Lower Limb Strength, Power and Performance in Footballers
Brief Title: Accentuated Eccentric Loading Versus Flywheel Exercises in Footballers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0454
Record Dates: First submitted 2025-05-15; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Sports Physical Therapy
Keywords: Agility; Clinical trials; Football; Power; Randomized; Strength training

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Accentuated Eccentric Loading training
  Interventions: Other: Accentuated Eccentric Loading training
- Group B (Experimental): Flywheel exercises
  Interventions: Other: Flywheel exercises

INTERVENTIONS:
Other: Accentuated Eccentric Loading training — 18 particpants will train in AEL group for three days a week for eight weeks and each session will take about 60-75 minutes, focusing on eccentric exercises like back squats, leg press, and hip thrusts at 90% 1RM intensity. Sessions, supervised by coaches, include free weight and weight machine exercises. Performance tests (20m sprint, T-agility, broad jump, 1RM assessments) will evaluate progress at the study's start and end.
  Arms: Group A
Other: Flywheel exercises — 18 particpants will train in FW group for three days a week for eight weeks and each session will take about 60-75 minutes, incorporating compound movements, Flywheel exercises (squats, sprints, jumps), and relevant free weight and weight machine exercises. Supervised sessions maintain consistent parameters. Performance tests (20m speed, T-agility, broad jump, 1RM assessments) will measure improvements at study start and end for evaluation.
  Arms: Group B

SUMMARY:
In the field of football, the essence of the lower limb strength, power and general performance is greatly valued by any player who wants to perform exceptionally well in both the acceleration, jumping and general agility. Conventional strengthening techniques have always been basic and recent strategies such as the Accentuated Eccentric Loading (AEL) and Flywheel (FW) have been considered as the inventions. AEL increases the muscle contraction during the eccentric phase of exercises and therefore improves hypertrophy and strength. On the other hand, FW uses leverage kinetic energy to oppose, thus, promotes muscle contractions and changes constantly. There is different training modalities that can be applied during training sessions or in prepare to a particular event such as football. Thus, it is essential to compare the applicability of those modalities in training football players. This study design will be Randomized clinical trial. Thirty-six male age 18-21 years who consistently play football and participate in resistance training from previous one year will randomly assigned to the two different exercise protocol i.e. Accentuated eccentric loading and Flywheel. The participants will undergo training program for total of 8 weeks. These two groups will exercise three days in a week and each session will take about 60-75 minutes. In this study researcher will use Back Squat and Leg Press for lower limb strength. Hip thrusts and Broad Jump for lower limb power. Free weights or Weight Machines, 20- meter sprint test and Agility T-test to measure performance of footballers. Data will be analyzed using SPSS version 25.

DETAILED DESCRIPTION:
The objective of this study is to compare the impact of Accentuated Eccentric Loading and Flywheel exercises on lower limb strength, power and performance in Football Players.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-21 years
* Only male participants.
* At least two years of resistance training experience
* Consistent participation in football and resistance training for at least one year prior to the study

Exclusion Criteria:

* Neuromuscular or musculoskeletal disorders.
* Participants have undergone any kind of surgery.
* Systematic illness: diabetic, hypertension, Trauma or accident history

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 36 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Back Squat | 8 weeks
  Back squats compose muscular strength of lower limbs and hence, they were performed at a load of 90% of 1 RM. They recruit the quadriceps, hamstrings, gluteal muscles and the lower back skeletal muscles. It can be concluded that back squat as a measure of maximal strength is reliable and valid especially in athletic subjects such as football players. Cronbach alpha is significant in strength assessment in sports using back squats; test-retest reliability ICC equals 0. 97 and construct validity has been discovered in existing works.
Hip Thrusts | 8 weeks
  At 90% 1RM hip thrust with the barbell aims at the gluteal muscles and plays an essential role in the improvement of hip extension power needed profoundly in sprinting and jumping in football. This exercise has been proven to help in enhancing hip strength as well as sprint performance; meanwhile, the reliability coefficient of the test in measuring maximal strength in athletes was very high (ICC = 0. 94). The hip thrust's focus on the posterior chain renders it a measure of lower limb strength that is directly applicable to football performance.
Broad Jump | 8 weeks
  The broad jump is a test that is frequently used in lower body power, which tracks the force thatan individual athlete is able to produce quickly. This exercise is quite pertinent for football players since it replicates the kind of movements involved in football. The broad jump has shown test-retest reliability of Internal Consistency Coefficient, ICC= 0. 95 and construct validity in determining lower body power of athletes. It is easy to administer, sensitive and reliable and thus widely accepted as a standard measure in athletic ability assessment.
Leg Press Machine | 8 weeks
  The leg-press equipment is used perform unilateral leg-press exercise to determine 1-RM strength and the maximal voluntary isometric contraction (MVIC). This exercise focuses on the quadriceps, hamstrings, and glutes by comparatively giving a controlled situation to determine lower limb force. In correlating maximal strength in the context of the leg press, previous studies have found very high to almost perfect reliability (ICC = 0. 96) as well as validity in populations that demand accurate determination of unilateral leg strength.
Agility T-test | 8 weeks
  Agility T-test checks how quickly players can change direction and control their body. Players start by sprinting forward, go around a cone, weave through middle cones to the top, turn, weave back through, circle another cone, and sprint to the finish. This tool reliability showed a highICC in almost all studies.
20 Meter Sprint test | 8 weeks
  The 20m sprint test assesses speed over a greater distance compared to the 10m sprint test. Studies have demonstrated that the 20m Sprint Test maintains validity and reliability when performed using electronic timing gates.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Dring Stadium, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaabene H, Markov A, Prieske O, Moran J, Behrens M, Negra Y, Ramirez-Campillo R, Koch U, Mkaouer B. Effect of Flywheel versus Traditional Resistance Training on Change of Direction Performance in Male Athletes: A Systematic Review with Meta-Analysis. Int J Environ Res Public Health. 2022 Jun 9;19(12):7061. doi: 10.3390/ijerph19127061. PMID 35742311
- [Background] Nuzzo JL, Pinto MD, Nosaka K. Connective Adaptive Resistance Exercise (CARE) Machines for Accentuated Eccentric and Eccentric-Only Exercise: Introduction to an Emerging Concept. Sports Med. 2023 Jul;53(7):1287-1300. doi: 10.1007/s40279-023-01842-z. Epub 2023 Apr 25. PMID 37097413
- [Background] Godwin MS, Fearnett T, Newman MA. The Potentiating Response to Accentuated Eccentric Loading in Professional Football Players. Sports (Basel). 2021 Nov 26;9(12):160. doi: 10.3390/sports9120160. PMID 34941798
- [Background] Weng Y, Liu H, Ruan T, Yang W, Wei H, Cui Y, Ho IMK, Li Q. Effects of flywheel resistance training on the running economy of young male well-trained distance runners. Front Physiol. 2022 Dec 8;13:1060640. doi: 10.3389/fphys.2022.1060640. eCollection 2022. PMID 36569754
- [Background] Stojanovic MDM, Mikic M, Drid P, Calleja-Gonzalez J, Maksimovic N, Belegisanin B, Sekulovic V. Greater Power but Not Strength Gains Using Flywheel Versus Equivolumed Traditional Strength Training in Junior Basketball Players. Int J Environ Res Public Health. 2021 Jan 29;18(3):1181. doi: 10.3390/ijerph18031181. PMID 33572738
- [Background] Negra Y, Chaabene H, Sammoud S, Prieske O, Moran J, Ramirez-Campillo R, Nejmaoui A, Granacher U. The Increased Effectiveness of Loaded Versus Unloaded Plyometric Jump Training in Improving Muscle Power, Speed, Change of Direction, and Kicking-Distance Performance in Prepubertal Male Soccer Players. Int J Sports Physiol Perform. 2020 Feb 1;15(2):189-195. doi: 10.1123/ijspp.2018-0866. Epub 2019 Oct 15. PMID 31094246
- [Background] Sagelv EH, Pedersen S, Nilsen LPR, Casolo A, Welde B, Randers MB, Pettersen SA. Flywheel squats versus free weight high load squats for improving high velocity movements in football. A randomized controlled trial. BMC Sports Sci Med Rehabil. 2020 Oct 2;12:61. doi: 10.1186/s13102-020-00210-y. eCollection 2020. PMID 33024564
- [Background] di Cagno A, Iuliano E, Buonsenso A, Giombini A, Di Martino G, Parisi A, Calcagno G, Fiorilli G. Effects of Accentuated Eccentric Training vs Plyometric Training on Performance of Young Elite Fencers. J Sports Sci Med. 2020 Nov 19;19(4):703-713. eCollection 2020 Dec. PMID 33239944
- [Background] Wang J, Zhang Q, Chen W, Fu H, Zhang M, Fan Y. The effect of flywheel complex training with eccentric-overload on muscular adaptation in elite female volleyball players. PeerJ. 2024 Mar 21;12:e17079. doi: 10.7717/peerj.17079. eCollection 2024. PMID 38525282
- [Background] Oliver JL, Ramachandran AK, Singh U, Ramirez-Campillo R, Lloyd RS. The Effects of Strength, Plyometric and Combined Training on Strength, Power and Speed Characteristics in High-Level, Highly Trained Male Youth Soccer Players: A Systematic Review and Meta-Analysis. Sports Med. 2024 Mar;54(3):623-643. doi: 10.1007/s40279-023-01944-8. Epub 2023 Oct 28. PMID 37897637
- [Background] Armitage M, McErlain-Naylor SA, Devereux G, Beato M, Buckthorpe M. On-field rehabilitation in football: Current knowledge, applications and future directions. Front Sports Act Living. 2022 Dec 5;4:970152. doi: 10.3389/fspor.2022.970152. eCollection 2022. No abstract available. PMID 36544545
- [Background] Yuan S, Lu Z, Tan S, Zhang Z, Jing S, Liu H, Zhou Z, Bao D. Comparison of six-week flywheel and traditional resistance training on deceleration and dynamic balance in elite badminton players. Front Physiol. 2025 Feb 25;16:1491661. doi: 10.3389/fphys.2025.1491661. eCollection 2025. PMID 40070459
- [Background] Beato M, Dello Iacono A. Implementing Flywheel (Isoinertial) Exercise in Strength Training: Current Evidence, Practical Recommendations, and Future Directions. Front Physiol. 2020 Jun 3;11:569. doi: 10.3389/fphys.2020.00569. eCollection 2020. No abstract available. PMID 32581845
- [Background] Maroto-Izquierdo S, Martin-Rivera F, Nosaka K, Beato M, Gonzalez-Gallego J, de Paz JA. Effects of submaximal and supramaximal accentuated eccentric loading on mass and function. Front Physiol. 2023 Jun 28;14:1176835. doi: 10.3389/fphys.2023.1176835. eCollection 2023. PMID 37449014
- [Background] Perna P, de Keijzer KL, Beato M. Flywheel resistance training in football: a useful rehabilitation tool for practitioners. Front Sports Act Living. 2024 Jul 5;6:1434995. doi: 10.3389/fspor.2024.1434995. eCollection 2024. No abstract available. PMID 39036368